CLINICAL TRIAL: NCT02718040
Title: A Multi-Center Study to Evaluate the Perception of Facial Expressions Following Correction of Wrinkles and Folds in the Lower Face Using Emervel® Classic Lidocaine and Emervel® Deep Lidocaine
Brief Title: Emervel for the Correction of Lower Face Wrinkles & Folds
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLI.04.SPR.US10345
Record Dates: First submitted 2016-03-16; First posted 2016-03-24 (Estimated); Results first posted 2018-09-25 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2018-09

CONDITIONS: Nasolabial Folds; Marionette Lines; Wrinkles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Emervel Treatment Group (Experimental): Eligible subjects received bilateral treatment of Nasolabial Folds (NLFs) and Marionette Lines (MLs) with Emervel Classic and/or Emervel Deep
  Interventions: Device: Emervel Classic and/or Deep Treatment Group

INTERVENTIONS:
Device: Emervel Classic and/or Deep Treatment Group — Severity of Wrinkle Severity treated by product type:
  Emervel Classic:
  Nasolabial Folds (NLFs): Wrinkle Severity Rating Scale (WSRS) = 2/2, 2/3 or 3/3; Marionette Lines (MLs): Wrinkle Assessment Scale (WAS) = 2/2, 2/3 or 3/3
  Emervel Deep Nasolabial Folds (NLFs): Wrinkle Severity Rating Scale (WSRS) = 3/3, 3/4 or 4/4; Marionette Lines (MLs): Wrinkle Assessment Scale (WAS) = 3/3, 3/4 or 4/4
  Both products may be used in the same subject, but only in different anatomic locations. The same study product should be used within the same wrinkle or fold type (e.g., left and right NLFs treated with the same product)

SUMMARY:
This study is designed to

1. evaluate the naturalness of facial expressions in motion (2D video images), by treating investigator assessment
2. evaluate naturalness of facial expressions (photographs), by treating investigator assessment
3. evaluate perceived attractiveness and age of subject (2D videos), by treating investigator assessment
4. evaluate aesthetic improvement, by subject and treating investigator assessments
5. evaluate subject satisfaction
6. evaluate nasolabial fold (NLF) severity, by treating investigator assessment
7. evaluate marionette lines (MLs) severity, by treating investigator assessment
8. evaluate dynamic facial strain in animation using 3D digital photogrammetric analysis
9. evaluate all adverse events reported during the study.

ELIGIBILITY:
Key Inclusion Criteria:

1. Seeking correction of bilateral NLFs: severe (i.e., bilateral WSRS = 3-4) or moderate (i.e., bilateral WSRS = 2-3) AND bilateral MLs: severe (i.e., WAS = 3-4) or moderate (i.e., WAS = 2-3).
2. Subjects of childbearing potential who agree to use medically accepted methods of contraception during the study and for 30 days following study completion.
3. Intent to undergo optimal correction of bilateral NLFs and MLs. Optimal correction is defined as the best possible aesthetic outcome as agreed to by the treating investigator and subject.

Key Exclusion Criteria:

1. Subject who presents with a severity of wrinkles or folds that require other treatments, e.g. laser treatment, chemical peeling, to achieve optimal correction.
2. Previous facial surgery, including aesthetic facial surgical therapy, liposuction or tattoo, in the treatment area.
3. Previous tissue augmenting therapy or contouring with permanent or non-permanent filler or fat-injection in the facial area.
4. Previous tissue revitalization treatment with neurotoxin in the facial area within 6 months before treatment.
5. Known/previous allergy or hypersensitivity to any injectable hyaluronic acid (HA) gel.
6. Known/previous allergy or hypersensitivity to local anaesthetics, e.g. lidocaine or other amide-type anaesthetics.
7. Known/previous allergy or hypersensitivity to gram-positive bacterial proteins.
8. Any medical condition that, in the opinion of the treating investigator, would make the subject unsuitable for inclusion (e.g. a chronic, relapsing or hereditary disease that may interfere with the outcome of the study).
9. Other condition preventing the subject from entering the study in the treating investigator's opinion, e.g. subjects not likely to avoid other facial cosmetic treatments, subjects anticipated to be unreliable, unavailable or incapable of understanding the study assessments or having unrealistic expectations of the treatment result.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Mashburn, Study Director — Galderma Laboratories

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Emervel Treatment Group: Eligible subjects received bilateral treatment of Nasolabial Folds (NLFs) and Marionette Lines (MLs) with Emervel Classic and/or Emervel Deep
  Emervel Classic and/or Deep Treatment Group: Severity of Wrinkle Severity treated by product type:
  Emervel Classic:
  Nasolabial Folds (NLFs): Wrinkle Severity Rating Scale (WSRS) = 2/2, 2/3 or 3/3; Marionette Lines (MLs): Wrinkle Assessment Scale (WAS) = 2/2, 2/3 or 3/3
  Emervel Deep Nasolabial Folds (NLFs): Wrinkle Severity Rating Scale (WSRS) = 3/3, 3/4 or 4/4; Marionette Lines (MLs): Wrinkle Assessment Scale (WAS) = 3/3, 3/4 or 4/4
  Both products may be used in the same subject, but only in different anatomic locations. The same study product should be used within the same wrinkle or fold type (e.g., left and right NLFs treated with the same product)
Period: Overall Study
Arm/Group | Emervel Treatment Group
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Emervel Treatment Group
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.0 (6.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Naturalness of Expression in Motion (2D Video)
Description: Proportion of subjects having at least maintained naturalness of expression in lower face (naturalness is maintained or enhanced) based on 2D video assessment at Day 42, by treating investigator
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Emervel Treatment Group
Number analyzed (Participants) | 30
Participants | 30

2. Secondary Outcome: Number of Subjects With Naturalness of Expression (Photographs)
Description: Proportion of subjects having at least maintained naturalness of facial expression based on photograph assessment at Day 42, by treating investigator
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Emervel Treatment Group
Number analyzed (Participants) | 30
Participants | 28

3. Secondary Outcome: Number of Subjects With Naturalness of Expression, Attractiveness AND Younger Appearance (2D Video)
Description: Proportion of subjects having at least maintained naturalness of expression in the lower face (naturalness is maintained or enhanced) AND attractiveness of the lower face is enhanced AND age of the lower face is younger, based on 2D video assessment at Day 42, by the treating investigator. The is a composite perception assessment; the proportion of subjects must meet all 3 criteria (maintain naturalness, maintain attractiveness, and appear younger in the lower face.
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Emervel Treatment Group
Number analyzed (Participants) | 30
Participants | 25

4. Secondary Outcome: Number of Subjects Reporting Global Improvement (Subject)
Description: Aesthetic improvement assessed by subject using the Global Aesthetic Improvement Scale (GAIS). The subject reported GAIS assessment was based on comparing Day 42 to baseline photographs with the following ratings: Very much improved, much improved, somewhat improved, no change, and worse. A clinically significant "global" improvement was defined as a score of improved, much improved, or very much improved.
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Emervel Treatment Group
Number analyzed (Participants) | 30
Participants | 30

5. Secondary Outcome: Number of Subjects Demonstrating Global Improvement (Treating Investigator)
Description: Aesthetic improvement assessed by treating investigator using the Global Aesthetic Improvement Scale (GAIS). The treating investigator reported GAIS assessment was based on comparing Day 42 to baseline photographs with the following ratings: Very much improved, much improved, somewhat improved, no change, and worse. A clinically significant "global" improvement was defined as a score of improved, much improved, or very much improved.
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Emervel Treatment Group
Number analyzed (Participants) | 30
Participants | 30

6. Secondary Outcome: Number of Subjects Reporting Satisfaction - The Overall Appearance of my Face Looks Natural
Description: Proportion of subjects responding with Strongly Agree or Agree. Subject reported satisfaction using a 5-point Likert scale questionnaire. Responses were 1-strongly disagree, 2-disagree, 3-neutral, 4-agree, and 5-strongly agree.
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Emervel Treatment Group
Number analyzed (Participants) | 30
Participants | 30

7. Secondary Outcome: Wrinkle Severity (Assess NLFs) - Proportion of Subjects With Bilateral Improvement of at Least 1 Grade in Wrinkle Severity
Description: Wrinkle severity assessed by treating investigator at Day 15/Touch and Day 42 using the Wrinkle Severity Rating Scale (WSRS). Assessments of both NLFs were graded according the following responses: 1-absent, 2-mild, 3-moderate, 4-severe, and 5-extreme. WSRS improvement from baseline included 1-grade improvement (reduction in WSRS) from baseline.
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Emervel Treatment Group
Number analyzed (Participants) | 30
Participants | 30

8. Secondary Outcome: Wrinkle Severity (Assess MLs) - Proportion of Subjects With Bilateral Improvement of at Least 1 Grade in Wrinkle Severity
Description: Wrinkle severity assessed by treating investigator at Day 15/Touch and Day 42 using the Wrinkle Assessment Scale (WAS). Assessments of both MLs were graded according the following responses: 0-no wrinkles, 1-just perceptible wrinkle, 2-shallow wrinkle, 3, moderately deep wrinkle, 4-deep wrinkle, well defined edges, 5-very deep wrinkle, redundant fold. WAS improvement from baseline included 1-grade improvement (reduction in WAS) from baseline.
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Emervel Treatment Group
Number analyzed (Participants) | 30
Participants | 30

9. Secondary Outcome: Mean Change in Dynamic Facial Strain (Stretch) at Day 42 Compared to Baseline - NLF Combined (Global Dynamic Assessment)
Description: Dynamic strain (stretch) results were analyzed using a Global Dynamic Assessment (GDA).The GDA averages strain (stretch) for the 4 predefined individual expressions, providing a global measure of dynamic strain (stretch), for a specific area of interest (ie, NLF). This value reflects the mean change in dynamic facial stretch at Day 42 compared to Baseline using 3D imaging.
Time Frame: baseline and 42 days
Measure: Mean (Standard Deviation); unit: Percent of Stretch
Arm/Group | Emervel Treatment Group
Number analyzed (Participants) | 30
Percent of Stretch | -1.836 (2.1025)

10. Secondary Outcome: Mean Change in Dynamic Facial Strain (Stretch) at Day 42 Compared to Baseline - ML Combined (Global Dynamic Assessment)
Description: Dynamic strain (stretch) results were analyzed using a Global Dynamic Assessment (GDA).The GDA averages strain (stretch) for the 4 predefined individual expressions, providing a global measure of dynamic strain (stretch), for a specific area of interest (ie, ML). This value reflects the mean change in dynamic facial stretch at Day 42 compared to Baseline using 3D imaging.
Time Frame: baseline and 42 days
Measure: Mean (Standard Deviation); unit: Percent of Stretch
Arm/Group | Emervel Treatment Group
Number analyzed (Participants) | 30
Percent of Stretch | -2.209 (2.8716)

ADVERSE EVENTS:
Time Frame: 42 days
Groups:
- Emervel Treatment Group: Eligible subjects receive bilateral treatment of Nasolabial Folds (NLFs) and Marionette Lines (MLs) with Emervel Classic and/or Emervel Deep
  Emervel Classic and/or Deep Treatment Group: Severity of Wrinkle Severity to be treated by product type:
  Emervel Classic:
  Nasolabial Folds (NLFs): Wrinkle Severity Rating Scale (WSRS) = 2/2, 2/3 or 3/3; Marionette Lines (MLs): Wrinkle Assessment Scale (WAS) = 2/2, 2/3 or 3/3
  Emervel Deep Nasolabial Folds (NLFs): Wrinkle Severity Rating Scale (WSRS) = 3/3, 3/4 or 4/4; Marionette Lines (MLs): Wrinkle Assessment Scale (WAS) = 3/3, 3/4 or 4/4
  Both products may be used in the same subject, but only in different anatomic locations. The same study product should be used within the same wrinkle or fold type (e.g., left and right NLFs treated with the same product)
Arm/Group | Emervel Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No